CLINICAL TRIAL: NCT03369613
Title: Transcranial Electrical Stimulation (tES) for the Treatment of Cervical Dystonia
Brief Title: Transcranial Electrical Stimulation for Cervical Dystonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-1322
Record Dates: First submitted 2017-11-29; First posted 2017-12-12 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Primary Cervical Dystonia
MeSH Terms: conditions — Cervical Dystonia, Primary | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- MRI - HC tDCS (Active Comparator): Healthy controls in Phase 1 transcranial electrical stimulation set to direct current
  Interventions: Device: transcranial electrical stimulation
- MRI - HC tACS (Active Comparator): Healthy controls in Phase 1- transcranial electrical stimulation set to alternating current
  Interventions: Device: transcranial electrical stimulation
- MRI - CD tCDS (Active Comparator): Cervical dystonia in Phase 1 transcranial electrical stimulation set to direct current
  Interventions: Device: transcranial electrical stimulation
- MRI - CD tACS (Active Comparator): Cervical dystonia in Phase 1 transcranial electrical stimulation set to alternating current
  Interventions: Device: transcranial electrical stimulation
- Phase II - Stim (Active Comparator): Cervical dystonia in Phase 2 transcranial electrical stimulation setting is active
  Interventions: Device: transcranial electrical stimulation
- Phase II - Sham (Sham Comparator): Cervical dystonia in Phase 2 transcranial electrical stimulation setting is sham
  Interventions: Device: transcranial electrical stimulation

INTERVENTIONS:
Device: transcranial electrical stimulation — The device is a Neoprene headcap that holds an array of padded electrodes close to the scalp to stimulate the underlying brain.

SUMMARY:
There are two phases.

Phase I: A single visit which includes a screening, clinical scales, and a MRI scan with simultaneous tES/sham tES in a randomized block design. Enrolls both Cervical Dystonia (CD) patients and healthy controls.

Phase II: 5 consecutive days of 30-90 min visits to campus for tES or sham tES. Transcranial magnetic stimulation (TMS) measures and clinical scales will also be included on Day 1 and Day 5 visits. Enrolls only CD patients.

DETAILED DESCRIPTION:
Phase I:

Enrolls both CD patients and healthy controls.

One approximately 3 hour visit which includes:

* a screening & neurological exam,
* clinical scales & questionnaires,
* a (approx.) 60 min MRI scan with simultaneous tES/sham tES in a randomized block design and EMG

Phase II:

Enrolls only CD patients.

Five consecutive days of study visits.

Day 1:

* TMS screening,
* repeated neurological assessment and clinical scales if >1 month since MRI visit
* 30 min TMS session with concurrent EMG
* 20 min tES or sham tES session

Days 2-4:

- 20 min tES or sham tES session

Day 5:

* 20 min tES or sham tES session
* 30 min TMS session with concurrent EMG
* repeated neurological assessment and clinical scales

ELIGIBILITY:
Primary Cervical Dystonia

Inclusion Criteria:

* Right-handed
* On a stable dose of all medications used to treat dystonia for the month previous to enrollment
* No botox injections in the 10 weeks previous to enrollment

Exclusion Criteria:

* Any contraindication to MRI scanning, tES, or TMS (e.g pregnancy, history of seizures, significant systemic medical conditions, untreated psychiatric or neurological conditions)
* Evidence on neurological exam of any potentially confounding neurological disorder
* Evidence of significant cognitive impairment
* Patients with dystonia symptoms beginning prior to the age of 18 will be excluded
* Patients with secondary dystonia resulting from medications or that are part of another neurological disorder (e.g. Parkinson's disease) will be excluded
* Medication that might predispose the subject to seizures

Healthy Controls

Inclusion Criteria:

- Right-handed

Exclusion Criteria:

* Any contraindication to MRI scanning, tES, or TMS (e.g pregnancy, history of seizures, significant systemic medical conditions, untreated psychiatric or neurological conditions)
* Evidence on neurological exam of any potentially confounding neurological disorder
* Evidence of significant cognitive impairment
* Medication that might predispose the subject to seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Phase I: A change in brain functional connectivity in primary cervical dystonia | Day 1
  A change in mean functional connectivity between the pallidum and putamen during a resting state in CD patients during inhibitory tACS targeting the sensorimotor network.
Phase II: Improvement in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) score | Day 1, Day 5
  A change in TWSTRS scores following five daily sessions of inhibitory tACS.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Berman, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States